CLINICAL TRIAL: NCT00761371
Title: Exploratory Evaluation of Imiquimod 5% Cream in the Treatment of External Genital or Perianal Warts in HIV+ Patients Treated With HAART (CD4+ ≥ 200 Cells mm3): An Open Labeled, Non-comparative Study
Brief Title: Imiquimod 5% Cream in the Treatment of External Genital or Perianal Warts in HIV+ Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Collaborators: ORION Sante (Unknown)
Responsible Party: Joachim Maus, MD / Director, Clinical Development, Meda Pharma GmbH & Co. KG
Organization: Viatris Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1456-IMIQ; X-03016-9359000001
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2015-04

CONDITIONS: Warts
Keywords: external genital and perianal warts
MeSH Terms: conditions — Warts | interventions — Imiquimod

ARMS (1):
- Imiquimod (Experimental): Imiquimod 5% cream
  Interventions: Drug: Imiquimod 5% cream

INTERVENTIONS:
Drug: Imiquimod 5% cream — Subjects were treated with imiquimod (one sachet/20 cm2), three applications per week, for up to 16 weeks, or fewer in the case of total clearance of initial warts. At the visit at the end of treatment, a second scraping of the lesion area was carried out to determine the sub-type of HPV.

SUMMARY:
Imiquimod 5% cream in the treatment of external genital or perianal warts in HIV+ patients

DETAILED DESCRIPTION:
To evaluate the percentage of HIV+ subjects successfully treated with HAART, with total clearance (100%) of baseline external genital or perianal warts within 16 weeks of treatment with imiquimod 5% cream.

ELIGIBILITY:
Inclusion Criteria:

1. Subject able to understand and willing to give written informed consent.
2. Subject ≥ 18 and < 70 years of age.
3. Male or female with an HIV infection documented by serology (enzyme linked immunoabsorbent assay (ELISA)), Western Blot assay, or HIV viral load.
4. Treated with HAART for at least six months and compliant with the treatment.
5. Evidence of efficacy of HAART: total CD4+ lymphocyte counts of ≥ 200 cells/mm3 AND plasma HIV RNA level < 104 RNA copies/mL within four weeks prior to the Treatment Initiation Visit.
6. Presence of at least one visible genital or perianal wart as determined by clinical diagnosis.
7. Total wart area > 10 mm2 and ≤ 4000 mm2 (diameter > 0.4 cm and ≤ 7.1 cm)
8. Karnofsky Performance Status ≥ 70 %.
9. Accepting to abstain from sexual intercourse when study drug is on the skin.
10. In case of a coexisting AIDS-defining illness, both this illness and any treatment being received for it must have been stable for the four weeks preceding enrolment in the trial.
11. If female and of childbearing potential, have negative urine pregnancy tests, and willing to use a medically acceptable method of contraception during the 16-week treatment period. Subjects were considered to be of childbearing potential unless the uterus or both ovaries had been removed or they were two or more years postmenopausal. For this study, the following were considered to be acceptable methods of contraception:

    * Surgical sterilization, defined as tubal ligation of the subject or a vasectomy of the subject's partner if that subject is in a monogamous heterosexual relationship (at the Investigator's discretion)
    * Oral, injectable, or implantable contraceptives
    * Condoms (with spermicide)
    * Diaphragm/cervical cap (with spermicide)
    * Intrauterine devices (IUDs)
    * Complete abstinence (at the Investigator's discretion)

Exclusion Criteria:

1. Women pregnant or lactating;
2. Treatment within four weeks prior to the Treatment Initiation Visit and throughout the entire study with:

   * Any genital wart therapy, or Immunomodulators
   * Systemic antiviral drugs other than acyclovir, valacyclovir, or famcyclovir and other than HAART

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2002-08; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects with total clearance of initially treated external genital or perianal warts. | week 16

SECONDARY OUTCOMES:
Total clearance | week 16
Percentage of subjects with a partial reduction of initial wart area; | week 16
Time to achieve reduction in wart area; | week 16
Reduction in wart number | week 16
Appearance of new warts | week 16
Recurrence rate | week 16
HPV DNA | week 16
CD4+ lymphocyte and HIV RNA levels | week 16

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Saiag, MD, Prof., Principal Investigator — Hospital Ambroise Pare, Department of Dermatology
Locations (17):
- Belgium (4):
  - Départment de Gynécologie-Obstétrique CHU Saint-Pierre, Brussels
  - Service de Dermatologie CHU Saint-Pierre, Brussels
  - Service Dermatologie C.H. François Rabelais (César de Paepe), Brussels
  - Service de Dermatologie Hôpital Erasme, Brussels
- France (13):
  - Service de Dermatologie et Vénéréologie Hôpital Saint Jacques, Besançon
  - Cabinet Médical, Bordeaux
  - Service de Dermatologie, Hôpital Ambroise Paré, Boulogne-Billancourt
  - Service de Maladies Infectieuses Hôpital de la Conception, Marseille
  - Service de Dermatologie Hôtel Dieu, Nantes
  - Service de Dermatologie Hôpital de l'Archet II, Nice
  - Service Dermatologie Hopital COCHIN - Pavillon Tarnier, Paris
  - Cabinet Médical, Paris
  - Institut Alfred Fournier, Paris
  - Service de Dermatologie Groupe Hospitalier Bichat Claude Bernard, Paris
  - Service de Dermatologie Hopital Tenon, Paris
  - Service de Dermatologie Groupe Hospitalier La Grave, Toulouse
  - Service de Dermatologie Centre Hospitalier de Valence, Valence

REFERENCES:
- [Derived] Saiag P, Bauhofer A, Bouscarat F, Aquilina C, Ortonne JP, Dupin N, Mougin C. Imiquimod 5% cream for external genital or perianal warts in human immunodeficiency virus-positive patients treated with highly active antiretroviral therapy: an open-label, noncomparative study. Br J Dermatol. 2009 Oct;161(4):904-9. doi: 10.1111/j.1365-2133.2009.09210.x. Epub 2009 May 15. PMID 19466962